CLINICAL TRIAL: NCT00128869
Title: Comparison of the Effectiveness of Mobilization and Manipulation of the Thoracic Spine in Patients With Mechanical Neck Pain: A Randomized Clinical Trial
Brief Title: Comparison of the Effectiveness of Mobilization and Manipulation of the Thoracic Spine in Patients With Mechanical Neck Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Newton-Wellesley Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NO5-368
Record Dates: First submitted 2005-08-09; First posted 2005-08-10 (Estimated); Last update posted 2008-05-13 (Estimated); Status verified 2008-05

CONDITIONS: Neck Pain
Keywords: Manipulation; Mobilization; Neck Pain; Physical Therapy
MeSH Terms: conditions — Neck Pain

INTERVENTIONS:
Procedure: spine mobilizations
Procedure: spine manipulations

SUMMARY:
This study aims to compare whether or not there is a difference in the effectiveness of upper back (thoracic spine) mobilizations versus manipulations used in a population of patients with mechanical neck pain. The investigators hypothesize that patients receiving a manipulative technique will experience better outcomes than patients receiving the mobilization techniques and these results will be evident at a 48-hour follow-up.

DETAILED DESCRIPTION:
Patients with mechanical neck pain who meet the study's inclusion criteria, who do not meet the study's exclusion criteria will be offered an opportunity to participate in this study. They will be issued an informed consent detailing the study and will have time to decide whether or not to participate. Once they have enlisted in the study they will complete forms to assess their current functional level. The investigator will then perform a standard clinical exam on the upper quarter to include a comprehensive subjective examination, upper extremity strength, reflexes, sensory assessment, cervical range of motion, thoracic range of motion and pain assessment. Once the above data have been collected and the patient has met the criteria for the study, a second investigator will then choose a randomized and sealed envelope which will indicate the treatment to be performed. The patient will either receive mobilization or manipulation to the thoracic spine. Mobilizations will be performed in prone over the spinous processes of T1-T6. Each one will be performed for 30 seconds each with force directed posterioanterior. The manipulation will be performed in supine with the patient's arms crossed over his/her chest. The therapist will pull the patient's arms downward to create spinal flexion down to the level where the manipulation will occur. The therapist's manipulative hand will stabilize the lower vertebrae of the motion segment and his/her body will be used to push down through the patient's arms to perform a high velocity, low amplitude thrust of the superior vertebrae. The manipulation will first be attempted in the upper thoracic spine; if a cavitation is heard on the first attempt he/she will move onto the middle thoracic area. If a cavitation is not heard he/she will attempt a second time before moving on to the next area. Both areas will receive a maximum of two attempts. Once the manipulation or mobilization is performed the patient will be assigned one home exercise which includes rotation of the cervical spine in both directions for 10 reps, 3-4 times per day. The patient will return within 48 hours for final data collection which will include a global rating of change scale completed both by the therapist and the patient, pain diagram and scale, neck disability index, cervical and thoracic range of motion measurements, and a side effects questionnaire. The patient will then be discharged from the study and will continue with physical therapy as deemed appropriate at the time of examination.

ELIGIBILITY:
Inclusion Criteria:

* Primary complaint of neck pain with duration of symptoms greater than 4 weeks
* Age between 18-60 years old

Exclusion Criteria:

* Red flags from the medical neck screening questionnaire to include tumor, fracture, metabolic disease, rheumatoid arthritis (RA), osteoporosis, prolonged history of steroid use.
* History of whiplash injury
* Diagnosis of cervical spinal stenosis
* Bilateral upper extremity symptoms
* Evidence of central nervous system involvement to include hyperreflexia, sensory disturbances in the hand, intrinsic muscle wasting of the hands, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, presence of pathological reflexes
* Two or more positive neurological signs consistent with nerve root compression to include muscle weakness involving a major muscle group of the upper extremity; diminished upper extremity muscle stretch reflex; diminished or absent sensation to pinprick in any upper extremity dermatome.
* Prior surgery to the neck or thoracic spine
* Pending legal action regarding neck pain

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2005-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Pain Diagram and Scale
Neck Disability Scale
Global Rating of Change Scale

SECONDARY OUTCOMES:
Side Effects Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Glynn, DPT, OCS, Principal Investigator — Newton-Wellesley Hospital
Locations (4):
- United States (4):
  - Sharp Rees-Stealy Medical Group, San Diego, California
  - Centennial Physical Therapy-Colorado Sport and Spine Centers, Colorado Springs, Colorado
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Groves Physical Therapy, Brooklyn Center, Minnesota

REFERENCES:
- [Background] Norlander S, Aste-Norlander U, Nordgren B, Sahlstedt B. Mobility in the cervico-thoracic motion segment: an indicative factor of musculo-skeletal neck-shoulder pain. Scand J Rehabil Med. 1996 Dec;28(4):183-92. PMID 9122645
- [Background] Norlander S, Gustavsson BA, Lindell J, Nordgren B. Reduced mobility in the cervico-thoracic motion segment--a risk factor for musculoskeletal neck-shoulder pain: a two-year prospective follow-up study. Scand J Rehabil Med. 1997 Sep;29(3):167-74. PMID 9271151
- [Background] Norlander S, Nordgren B. Clinical symptoms related to musculoskeletal neck-shoulder pain and mobility in the cervico-thoracic spine. Scand J Rehabil Med. 1998 Dec;30(4):243-51. doi: 10.1080/003655098443995. PMID 9825389
- [Result] Flynn TW, Wainner RS, Whitman JM. Immediate effects of thoracic spine manipulation on cervical range of motion and pain. Journal or Manual and Manipulative Therapy. 9(3), 164-171. 2001
- [Result] Cleland JA, Childs JD, McRae M, Palmer JA, Stowell T. Immediate effects of thoracic manipulation in patients with neck pain: a randomized clinical trial. Man Ther. 2005 May;10(2):127-35. doi: 10.1016/j.math.2004.08.005. PMID 15922233
- See also: American Physical Therapy Association Web Site — http://www.APTA.org
- See also: American Academy of Orthopaedic Manual Physical Therapy web site — http://aaompt.org